CLINICAL TRIAL: NCT02087735
Title: Measurement of Urinary Catabolites of the Proanthocyanidines (PACs) in Healthy Young Women as Biomarkers of Consumption of Cranberry Extracts.
Brief Title: Measurement of Urinary Catabolites of PACs as Biomarkers of Consumption of Cranberry Extracts
Acronym: CUPACS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Sylvie Dodin, Sylvie Dodin, MD, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PACS-2013-SD
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Tract Infections
Keywords: Cranberry; Proanthocyanidins; Urinary catabolites
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cranberry extract 1 (Experimental): One capsule with a proanthocyanidin standardized cranberry extract of 36 mg and one capsule of placebo cranberry extract.
  Interventions: Dietary Supplement: Cranberry extract
- cranberry extract 2. (Experimental): Two capsules with a proanthocyanidin standardized cranberry extract of 36 mg.
  Interventions: Dietary Supplement: Cranberry extract
- cranberry extract 3. (Placebo Comparator): Two capsules with a proanthocyanidin standardized cranberry extract of 2 mg.
  Interventions: Dietary Supplement: Cranberry extract

INTERVENTIONS:
Dietary Supplement: Cranberry extract — The aim of this pilot study is to evaluate the urinary catabolites of PACs as a biomarker of consumption of cranberry extracts within 9 hours of intercourse. Once a week, for 3 weeks, the women will receive a sequence of 3 different cranberry extracts (72 mg, 36 mg and 2mg (placebo)). The participant will have to collect its urine for a period of 9 hours in 3 different containers (one different container for 3 hours).

SUMMARY:
The purpose of this cross over pilot study is to investigate the urinary catabolites of Proanthocyanidines (PACs) as biomarkers of cranberry extracts in healthy young women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women.
* 18 to 40 years.

Exclusion Criteria:

* No internet access.
* No refrigerator access during the 9 hours of sample collection.
* Women who had or expect to take antibiotic.
* Women who had or expect to take cranberries, blueberries or bilberries in the form of berries, juice or extracts.
* Women who had or expect to take dark chocolate.
* Women who had personal history of acute or chronic renal failure.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Urinary catabolites of PACs | within 9 hours following the intake of cranberry extracts

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Dodin, MD, Principal Investigator — Laval University
Locations (1):
- Laval University, Department of Medecine, Institut sur la nutrition et les aliments fonctionnels (INAF)., Québec, Quebec, Canada